CLINICAL TRIAL: NCT03151941
Title: A Feasibility Study Monitoring the Respiratory Status of Participants Receiving or Scheduled to Receive Intrathecal Baclofen (ITB)
Brief Title: Respiratory Monitoring of Intrathecal Baclofen- a Feasibility Study
Status: Completed | Type: Observational
Sponsor: Solent NHS Trust (Other Government)
Responsible Party: Sponsor
Other Study IDs: 1
Record Dates: First submitted 2017-03-13; First posted 2017-05-12 (Actual); Last update posted 2017-10-10 (Actual); Status verified 2017-10

CONDITIONS: Intrathecal Baclofen; Multiple Sclerosis; Respiratory System; Cerebral Palsy
MeSH Terms: conditions — Multiple Sclerosis; Cerebral Palsy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The methodology is a feasibility study to determine the feasibility of assessing people in the community with a neurological condition before proceeding towards a full powered community trial evaluating the influence of intrathecal baclofen.

DETAILED DESCRIPTION:
The purpose of this proposed research will evaluate a feasible method to assess the respiratory status of people with neurological conditions receiving or scheduled to receive Intrathecal Baclofen. The use of Intrathecal Baclofen to manage severe spasticity is a developing treatment option with a limited research base, particularly when evaluating the influence of intrathecal baclofen on the respiratory system. The proposed research is derived from clinical practice and involves joint collaboration between clinical team, research professionals and patients.

In order for the study to evaluate the influence of Intrathecal baclofen has on the respiratory system, the proposed research will need to develop and evaluate a method of assessing people in the community ensuring it's feasible for people with neurological conditions. Prior to implementing a full powered community trial to evaluate the influence of intrathecal baclofen on people with neurological conditions.

ELIGIBILITY:
Inclusion Criteria:

* -Adults over the age of 18
* A person who is able to provide consent or a family member/ close friend who is able to assent on behalf of the participant
* A person or a family member/ close friend who is able to understand English (understand written English and spoken instructions)
* A person currently receiving Intrathecal Baclofen or is scheduled to receive Intrathecal Baclofen (awaiting fitting of pump) therapy to manage spasticity
* A patient of the Solent/ University Hospitals Southampton NHS Foundation Trust Intrathecal baclofen service

Exclusion Criteria:

* -Pre-existing use of overnight non-invasive ventilation (NIV) and is compliant with NIV treatment
* A person who is unable to consent to the study and does not have a family/ close person to assent
* The study will exclude a person who is unable to independently remove the polysomnography and is also without supervision from another person (carer or partner) during the night. This ensures the participant is able to take off the polysomnography (or assisted by a carer) if it becomes uncomfortable and/or causes distress.

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People with Neurological conditions receiving or scheduled to receive intrathecal baclofen therapy.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2017-03-06 (Actual); Primary Completion 2017-08-31 (Actual); Study Completion 2017-08-31 (Actual)

PRIMARY OUTCOMES:
Overnight home polysomnography | 2 nights
  sleep study

SECONDARY OUTCOMES:
Sniff nasal inspiratory pressure Expiratory and inspiratory mouth pressures Cough peak flow Expanded disability status scale Epworth sleepiness scale Semi Structured interview | 2 nights
  Sniff nasal inspiratory pressure Expiratory and inspiratory mouth pressures Cough peak flow Expanded disability status scale Epworth sleepiness scale Semi Structured interview

CONTACTS AND LOCATIONS:
Overall Officials: Hayden Kirk, Principal Investigator — Solent NHS Trust
Locations (1):
- Solent NHS Trust, Portsmouth, Hampshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No